CLINICAL TRIAL: NCT07210073
Title: Video Assisted Education to Improve Blood Pressure Control in Ischemic Heart Disease Patients With Hypertension: Randomized Controlled Trial
Brief Title: Video Education to Improve Blood Pressure Control in Patients With Ischemic Heart Disease and Hypertension (V-EDUCATE)
Acronym: V-EDUCATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02-053
Record Dates: First submitted 2025-09-14; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-02

CONDITIONS: Hypertension (HTN); Ischemic Heart Disease
MeSH Terms: conditions — Hypertension; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video education (Experimental): Participants receive personalized video-based education developed using deepfake technology to replicate the patient's primary physician's voice, in addition to usual care.
  Interventions: Behavioral: Video Education
- Standard Care (Active Comparator): Participants receive standard treatment for ischemic heart disease and hypertension, without additional video-based education.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Video Education — Videos were created using deepfake technology, utilizing AI to replicate the voice of the patients' primary physician.
  Arms: Video education
Other: Control — Standard treatment
  Arms: Standard Care

SUMMARY:
We investigated whether video-based education using deepfake technology could improve blood pressure measurement adherence and medication adherence in patients with ischemic heart disease accompanied by hypertension.

DETAILED DESCRIPTION:
Hypertension is a major risk factor for recurrent cardiovascular events in patients with ischemic heart disease, yet adherence to home blood pressure monitoring and prescribed medications remains suboptimal. Personalized and engaging educational strategies may help to improve adherence behaviors in this population.

This randomized controlled trial investigates the effectiveness of a video-based educational program, developed with deepfake technology, to deliver individualized health information. Participants are randomly assigned to either the intervention group, which receives the video education in addition to usual care, or the control group, which receives usual care alone.

The primary outcomes are adherence to home blood pressure monitoring and medication adherence after one month. Secondary outcomes include changes in office and home blood pressure, as well as 24-hour ambulatory blood pressure monitoring. The results of this study may provide evidence for scalable, technology-assisted strategies to enhance adherence and improve blood pressure control in high-risk cardiovascular patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older, both male and female, with a history of hypertension or who have taken antihypertensive medication at least once, satisfying one or more of the following ischemic heart disease conditions (PCI, CABG, CAD >50% by CCT or CAG), or patients with a history of hypertension or currently taking antihypertensive medication.
* Individuals who have voluntarily provided written consent to participate in this clinical trial.

Exclusion Criteria:

* SBP < 90 mmHg or DBP < 50 mmHg
* Individuals intolerant to all antihypertensive medications
* Patients with heart failure due to other causes, Pregnant women, those suspected of being pregnant, or those who are breastfeeding
* Patients whom the investigator deems legally or mentally unfit to participate in the clinical trial
* Patients who have participated in another clinical study involving investigational drugs within 4 weeks prior to screening.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Adherence to Home Blood Pressure Monitoring (HBPM) | 4 weeks
  Proportion of days during the 30-day follow-up period in which participants recorded four BP measurements per day (two in the morning, two in the evening) using a validated home BP device (InBody BP170).
Medication Adherence Assessed by Pill Count | 4 weeks
  Proportion of prescribed antihypertensive medication doses taken during the 30-day follow-up period, assessed by pill counts at the follow-up visit.

SECONDARY OUTCOMES:
Change in Office Systolic Blood Pressure From Baseline to 4 Weeks | 4 weeks
  Mean change in systolic blood pressure (SBP) measured in clinic using a standardized sphygmomanometer at baseline and 4 weeks.
Change in Office Diastolic Blood Pressure From Baseline to 4 Weeks | 4 weeks
  Mean change in diastolic blood pressure (DBP) measured in clinic using a standardized sphygmomanometer at baseline and 4 weeks.
Difference in Mean Systolic Blood Pressure Between Home BP Monitoring and 24-Hour Ambulatory Monitoring | 4 weeks
  Difference between mean SBP values obtained from home BP monitoring (HBPM) and 24-hour ambulatory BP monitoring (ABPM).
Difference in Mean Diastolic Blood Pressure Between Home BP Monitoring and 24-Hour Ambulatory Monitoring | 4 weeks
  Difference between mean DBP values obtained from HBPM and ABPM.
Number of Antihypertensive Medications Prescribed Per Participant | 4 weeks
  Total number of prescribed antihypertensive medications per participant at baseline and at 4 weeks.
Distribution of Antihypertensive Medication Classes Used | 4 weeks
  Proportion of participants prescribed each class of antihypertensive medication (RAAS inhibitors, beta-blockers, calcium channel blockers, diuretics, etc.) at baseline and 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Keimyung University Dongsan Hospital, Daegu, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No